CLINICAL TRIAL: NCT04678297
Title: Role of Emotion Regulation on Low Back Pain Outcomes
Brief Title: Physical Activity Interventions To Heal Chronic Low Back Pain
Acronym: PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Crystal Park, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: H19-191; R01AT010555 (NIH)
Record Dates: First submitted 2020-12-17; First posted 2020-12-21 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain, physical activity, emotion regulation
MeSH Terms: conditions — Motor Activity; Emotional Regulation | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: We will employ blinding whenever possible. Assessments, evaluations, and data analysis will be conducted without knowledge of participants' assigned group. Study personnel will be blinded to the assigned condition of subjects when conducting data collection by using unique study identification numbers, by following a strict script to refrain from discussing participant activities, and by using different members of the study team to coordinate assigned condition activities and to collect data. De-identified data with codes for assigned condition will facilitate blinded data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical activity + emotion regulation group (Experimental): Participants randomized to the experimental group attend two group-based class sessions per week, each 1.25hours long, that are led by certified instructors who guide participants through various exercises. Participants are encouraged to practice the activities at home for 20 minutes each day.
  Interventions: Behavioral: Physical activity + emotion regulation intervention
- Physical activity control group (Active Comparator): Participants randomized to the control group attend two group-based class sessions per week, each 1.25hours long, that are led by trained therapists who guide participants through a series of stretching exercises. Participants are encouraged to practice the activities at home for 20 minutes each day.
  Interventions: Behavioral: Physical activity control intervention

INTERVENTIONS:
Behavioral: Physical activity + emotion regulation intervention — The intervention meet twice weekly for 12 weeks, 1.25 hrs./session. This intervention will be led by certified instructors trained in working with back pain patients. The instructor leads participants through a series of physical activity exercises at a slow-moderate pace. Participants will be asked to practice every day for 20 minutes to maximize the benefit of the intervention. Participants also receive a home practice manual containing some basic, safe postures that can be performed on days they are not attending the formal in-person sessions.
  Arms: Physical activity + emotion regulation group
Behavioral: Physical activity control intervention — The interventions meet twice weekly for 12 weeks, 1.25 hrs./session. This intervention is designed to require a similar amount of physical exertion. Classes involve conventional exercises appropriate for patients with CLBP, including a comprehensive set of exercises that stretch all the major muscle groups, with an emphasis on the trunk and legs. The intervention will include all 12 stretching exercises used in the exercise intervention of previous studies that have successfully used it in comparison to yoga, plus 3 additional stretches (hip internal rotators, hip adductors and hip flexion).Participants will be asked to practice every day for 20 minutes home as well. Printed handouts will be provided to facilitate home practice. In addition, a video demonstrating all the exercises will be provided to assist participants in practicing safely. Classes will be led by a licensed physical therapist who has previous experience leading exercise classes.
  Arms: Physical activity control group

SUMMARY:
This study will advance understanding on the mechanisms that mediate improved outcomes for chronic low back pain and provide specific directions for optimizing physical activity interventions for this population.

DETAILED DESCRIPTION:
In this study, participants with chronic low back pain will be randomized to receive a 12-week physical activity intervention (2 times per week with encouragement for home practice). The experimental condition will entail physical activity with components for strengthening emotion regulation skills, behaviors, and attitudes while the control condition will entail physical activity alone.

ELIGIBILITY:
Inclusion Criteria:

- Age > 18;

Report of low back pain >3 of last 6 months;

Willing to attend 12-weeks of yoga or stretching (twice per week);

Willing to complete 4 assessments;

English Literacy;

No changes in pain treatments in the past month;

Willing to not change pain treatments during study unless medically necessary;

Have not practiced yoga > 2x in the last 12 months;

Exclusion Criteria:

- back surgery within the last 1 year;

back pain due to specific systemic problem (e.g., lupus);

lower extremity weakness (motor strength 4/5 of the quads, gluts, hamstrings, EHL);

sciatica or (+) straight leg raise (SLR);

coexisting chronic pain problem (migraine headaches, fibromyalgia);

Serious or unstable psychiatric illness (e.g. psychosis, mania, history of suicide attempt);

major coexisting medical illness (e.g., cancer, COPD, morbid obesity);

Positive Romberg test (with or without sensory neuropathy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Emotion regulation abilities | Baseline and 6 weeks and 3 months and 6 months
  Difficulties in Emotion Regulation Scale - Change over time; range is 36-120, a higher score reflects less emotion regulation

SECONDARY OUTCOMES:
Pain severity/interference | Baseline and 6 weeks and 3 months and 6 months
  Brief Pain Inventory - Change over time; Brief Pain Inventory consists of 2 subscales: Pain Intensity (range from 0-40, higher scores are worse pain) and pain interference (range is 0-60, higher scores is greater interference)
Pain sensitization | Baseline and 6 weeks and 3 months and 6 months
  Quantitative sensory testing, Brief Pain Inventory - Change over time

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Park, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs Mansfield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that are part of National Institute of Health (NIH) designated common data elements collected during the trial, after de-identification have been submitted to NIH. Data can be accessed by directly submitting requests at that website.
Supporting Information: Study Protocol
Time Frame: Upon completion of all study analyses and publication of study results, anticipated to be December 2024
Access Criteria: Researchers who are actively conducting physical activity studies for participants with pain.

REFERENCES:
- [Derived] Starkweather AR, Xu W, Gnall KE, Emrich M, Garnsey CL, Magin ZE, Wu W, Fetta J, Groessl EJ, Park C. Testing Biological and Psychological Pathways of Emotion Regulation as a Primary Mechanism of Action in Yoga Interventions for Chronic Low Back Pain: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Mar 14;13:e56016. doi: 10.2196/56016. PMID 38483469